CLINICAL TRIAL: NCT01951924
Title: A European, Randomised, Double-blind, Active Comparator Controlled, Cross-over, Efficacy and Safety Study of a New 10% Ready To-use Liquid Human Intravenous Immunoglobulin (I10E) Versus Kiovig® in Patients With Multifocal Motor Neuropathy
Brief Title: LIME Study (LFB IVIg MMN Efficacy Study)
Acronym: LIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I10E-0901
Record Dates: First submitted 2013-09-20; First posted 2013-09-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Motor Neuron Disease
Keywords: Multifocal Motor Neuropathy
MeSH Terms: conditions — Motor Neuron Disease | interventions — gamma-Globulins; Administration, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: I10E then Kiovig® (Experimental): 1 g/kg for 1-3 days up to 2 g/kg for 2-5 days every 4 to 8 weeks (±7 days)
  Interventions: Drug: Biological : I10E (Human normal Immunoglobulin for intravenous administration 100mg/mL); Drug: Biological: Kiovig® (Human normal Immunoglobulin for intravenous administration 100mg/mL)
- Group B : Kiovig® then I10E (Experimental): 1 g/kg for 1-3 days up to 2 g/kg for 2-5 days every 4 to 8 weeks (±7 days)
  Interventions: Drug: Biological : I10E (Human normal Immunoglobulin for intravenous administration 100mg/mL); Drug: Biological: Kiovig® (Human normal Immunoglobulin for intravenous administration 100mg/mL)

INTERVENTIONS:
Drug: Biological : I10E (Human normal Immunoglobulin for intravenous administration 100mg/mL)
Drug: Biological: Kiovig® (Human normal Immunoglobulin for intravenous administration 100mg/mL)

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of I10E (LFB 10% ready-to-use liquid human intravenous immunoglobulin) compared to Kiovig® for the maintenance treatment of MMN in a randomized, double-blind, active comparator-controlled, cross-over trial.

DETAILED DESCRIPTION:
Multifocal motor neuropathy (MMN) is a chronic acquired, probably autoimmune, demyelinating, motor neuropathy. It is a rare disease, variable in its clinical features. The disease course is usually steadily progressive.

Intravenous immunoglobulin (IVIg) is the standard and the first line treatment for MMN. The Cochrane review of four randomized placebo-controlled studies showed a significant clinical improvement in muscle strength from IVIg in 78% of patients with MMN versus 4% with placebo but a non-significant improvement in disability (39% versus 11%) (van Schaik IN, 2005). However, IVIg treatment does not prevent a mild gradual decline in muscle strength which is probably due to ongoing axonal degeneration. In addition to its efficacy, IVIg is also a safe treatment with a positive benefit-risk ratio in MMN.

Muscle strength measured with the Modified Medical Research Council (MMRC 10) sum score as described in the study of Cats (Cats EA, 2008) including 20 movements i.e. 10 muscle groups of the upper and lower limbs on each side was selected as the primary endpoint. Other parameters of muscle strength such as measurement of grip strength by dynamometer - and functional disability will also be evaluated to reinforce the robustness of the study and substantiate the efficacy of I10E in MMN patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 18 to 80 years.
2. Written informed consent obtained prior to any study-related procedures.
3. Diagnosis of definite or probable MMN according to the EFNS/PNS Guideline 2010, First revision made by neuromuscular disease specialists with specific electrodiagnostic expertise.
4. Patients treated with a stable maintenance dose within 15% of any brand of IVIg (Kiovig® excluded) at 1 g/kg for 1-3 days up to 2 g/Kg for 2-5 days every 4 to 8 weeks (+/- 7 days), according to the EFNS/PNS Guideline 2010, First revision for at least 3 months prior to enrolment.
5. Covered by national health care insurance system if required by local regulations.

Exclusion Criteria:

1. Upper motor neuron, bulbar, cranial nerve or significant sensory deficit.
2. CSF protein >100 mg/dL (if available and done as part of a previous evaluation).
3. Any other ongoing disease that may cause neuropathy, such as toxin exposure, dietary difficency, uncontrolled diabetes, hyperthyroidism, cancer, systemic lupus erythematosus or other connective diseases, infection with HIV, hepatitis B virus (HBV), or hepatitis C (HCV), Lyme disease, multiple myeloma, Waldenström's macroglobulinemia, amyloid, and hereditary neuropathy.
4. BMI >= 40 kg/m2.
5. Known hypersensitivity to the active substance or to any of the excipients of I10E (glycine and polysorbate 80) or Kiovig(glycine).
6. Patient who have been treated with Kiovig shall not have received Kiovig during the last 6 months prior to enrolment.
7. History of IgA deficiency, except if the absence of anti-IgA antibodies is documented.
8. Protein-losing enteropathy characterised by serum protein levels <60 g/l and serum albumin levels <30 g/l or nephrotic syndrome characterised by proteinuria >=3.5 g/24 hours, serum protein levels <60 g/l and serum albumin levels <30 g/l.
9. History of cardiac insufficiency (New York Heart Association (NYHA) III/IV), uncontrolled cardiac arrythmia, unstable ischemic heart disease, or uncontrolled hypertension.
10. History of venous thrombo-embolic disease, myocardial infarction, or cerebrovascular accident.
11. Risk factor for blood hyperviscosity such as cryoglobulinemia or haematological malignancy with monoclonal gammopathy.
12. Glomerular filtration rate <80 ml/min/1.73m2 measured according to the Modified Diet in Renal Disease (MDRD) calculation.
13. Serum levels of AST, ALT >2 times upper limit of normal range.
14. Treatment within 12 months prior to screeening with immunomodulator or immunosuppressant agent (including but not limited to cyclophosphamide, cyclosporine, interferon-a, interferon-b 1a, anti-CD20, alemtuzumab, azathioprine, etanarcept, mycophenolate mofetil, methotrexate, haematopoietic stem cell transplantation).
15. Administration of another investigational product within the last month prior to inclusion.
16. Plasma exchange, blood products or derivatives administered with the last 3 months prior to screening.
17. Woman with positive results of pregnancy test or breast-feeding woman or woman of childbearing potential without an effective contraception.

    Effective contraception are injectible, patch or combined oestro-progestative or progestative contraceptives, Cooper T or levonorgest releasing intra-uterine devices, depot intramuscular medroxyprogesterone, subcutaneous progestative contraceptive implants, condoms or occlusive caps (diaphragm or cervical/vault caps) with spermicide, true abstinence (when this is in line with the preferred and usual lifestyle of the patient).
18. Any serious medical condition that would interfere with the clinical assessment of I10E or prevent the patient from complying with the protocol requirements.
19. Anticipated poor compliance of patient with study procedures during the 12 month duration of the study.
20. Drug or alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change between I10E and Kiovig® in the original MMRC 10 sum score described by Cats 2008 | at 6 months and 1 year

SECONDARY OUTCOMES:
Change between I10E and Kiovig® in: MMRC 10 new sum score (10 slightly different muscles on both sides) | at 6 months and 1 year
AEs observed and reported TAAEs (temporally associated AE) beginning at infusion or within 72H after infusion | from 49 to 56 weeks
Change between I10E and Kiovig® in : Rasch built MMRC sum score (Cats 2008) | at 6 months and 1 year
Change between I10E and Kiovig® in : INCAT: upper and lower limbs | at 6 months and 1 year
Change between I10E and Kiovig®: Grip strength | at 6 months and 1 year
Change between I10E and Kiovig® in: MMRC 14 sum score | at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc LEGER, MD, Principal Investigator — Hôpital de la Pitié Salpêtrière - Paris 75013
Locations (18):
- France (8):
  - CHU de Bordeaux -Hôpital Haut-Lévêque, Bordeaux
  - CHU Créteil - Groupe Hospitalier Henri Mondor, Créteil
  - CHRU Lille - Hôpital Roger Salengro, Lille
  - CHU de Lyon - Hôpital Pierre Wertheimer, Lyon
  - CHU de Marseille - Hôpital de La Timone, Marseille
  - CHU de Nice - Hôpital l'Archet, Nice
  - CHU Paris - Hôpital Pitié Salpétrière, Paris
  - CHU de Saint Etienne - Hôpital Nord, Saint-Etienne
- Italy (4):
  - Università di Genova - Ospedale San Martino, Genova
  - IRCCS Istituto Clinico Humanitas, Milan
  - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliero Universitaria San Giovanni Battista, Turin
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - Southampton General Hospital, Southampton